CLINICAL TRIAL: NCT01669694
Title: Women's Urology Center-Physical Therapy-Biomarkers Project
Brief Title: Pelvic Floor Physical Therapy-Biomarkers Project
Status: Completed | Type: Observational
Sponsor: Kenneth Peters, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2011-317
Record Dates: First submitted 2012-07-19; First posted 2012-08-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pelvic Pain
Keywords: Pelvic Pain; Pelvic Floor Physical Therapy; Biomarkers
MeSH Terms: conditions — Pelvic Pain | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with Pelvic Pain: Women with Pelvic Pain undergoing pelvic floor PT in the Beaumont Women's Urology Center
  Interventions: Other: Pelvic floor PT with biomarkers

INTERVENTIONS:
Other: Pelvic floor PT with biomarkers — Pelvic floor physical therapy and collection of urine for biomarker analysis.

SUMMARY:
This study is collecting serum and urine samples at various time points during pelvic floor physical therapy for women with pelvic pain.The biomarkers will be analyzed for cytokines and proteomics at various time points.

DETAILED DESCRIPTION:
Collection points will be baseline, and at the last PT visit.

ELIGIBILITY:
Inclusion Criteria:

* Women in the Beaumont Women's Urology Center who have pelvic pain and are starting pelvic floor PT in our center.

Exclusion Criteria:

* all others

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in the Beaumont Women's Urology Center who have pelvic pain and are starting pelvic floor PT in our center.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The change in biomarkers pre- and post-pelvic floor PT | pre- and post- pelvic floor PT
  Interim Analysis to be done as PI determines.

SECONDARY OUTCOMES:
Evaluation of biomarkers in relation to clinical findings | pre- and post- pelvic floor PT
  Clinical data and biomarkers will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Donna J Carrico, NP, MS, Principal Investigator — Corewell Health East; Kenneth Peters, MD, Study Chair — Corewell Health East
Locations (1):
- Beaumont Women's Urology Center, Royal Oak, Michigan, United States